CLINICAL TRIAL: NCT06413823
Title: Prevention and Treatment of Cardiovascular Disease: Protocol for the Assessment of Psychological, Neuropsychological Implications and Associated Disorders in Cardiology Patients
Brief Title: Prevention and Treatment of Cardiovascular Disease
Acronym: VPC
Status: Recruiting | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Irene Cappadona, Psychologist, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: 08/2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; neuropsychological; depression; anxiety; psychoeducation; dysphagia; caregiver; sleep disorders; altered pneumophonic coordination
MeSH Terms: conditions — Cardiovascular Diseases; Depression; Anxiety Disorders; Deglutition Disorders; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In view of the close interrelationship between the various organs and systems of the body, which cannot be examined in a parceled fashion but rather as an integrated system, this study aims to consider the potential risks associated with cardiovascular disease.

By identifying additional, often underestimated, altered functions that may affect the patient's quality of life and interfere with the performance of daily activities, this research study aims to evaluate the patient's functioning in an integrated manner to achieve a holistic view of the health and well-being of the patient and caregiver.

DETAILED DESCRIPTION:
The study design is observational and is planned to last approximately 24 months. The overall duration will be related to the time required for enrollment of all planned subjects, data analysis and publication of results.

The study aims to analyze and investigate the most common comorbidities in patients with cardiovascular disease. In addition, a specific focus will be devoted to the caregiver, who plays a key role for the cardiopathic patient.

In detail, the objectives of the project are:

1. Evaluate the connection between cardiovascular disease and cognitive deficits;
2. Evaluate the main psychopathologies related to cardiovascular diseases (anxiety, depression);
3. Evaluate conditions and disorders associated with cardiovascular diseases (dysphagia, pneumophonic coordination disorders, respiratory sleep disorders);
4. Evaluate the effectiveness of psychoeducational intervention;
5. Evaluate the impact of cardiovascular disease on the caregiver.

A minimum of 218 patients recruited from those afferent at the U.O.S.D. Cardiology with NICU P.O. "Piemonte" in Messina will participate in the survey. Statistical power analysis was performed using G*Power software for a linear regression test, assuming a slope (H1) of 0.2 with a significance level (α) of 0.05 and a power (1 - β) of 0.85. The primary outcome variable considered for the calculation is the result of the SF-12 (or SF-36) test as a summary index of the effectiveness of psychoeducation. The calculation indicated a sample of 218 subjects as adequate for the purpose of detecting the hypothesized effect.

Inclusion criteria:

* Age between 45 and 85 years;
* Confirmed diagnosis of cardiovascular disease;
* Presence of chronic cardiovascular disease;
* Absence of cognitive impairment or mild/moderate cognitive impairment (Mini Mental Score >26);
* Patient who has given informed consent personally or through Legal Representative.

Exclusion Criteria:

* Presence of severe psychiatric and neurological disorders.
* Presence of end-stage oncological disease.
* Severe visual impairment that cannot be corrected by dioptric lenses.

Each patient who is eligible for this study will be presented with the purpose of the study and will freely decide whether to join. Only after the patient, or his/her Legal Representative, has agreed to participate in the investigation and signed the informed consent, can the Investigator proceed with the planned activities, detailed below.

The patient's pathway should unfold as follows:

Each patient's clinical data will be shared from a database, accessible to study collaborators through previously assigned login credentials. After checking inclusion and exclusion criteria and signing informed consents, patients will be taken on.

1. Baseline Examination.

   * Verification of inclusion and exclusion criteria;
   * Collection of demographic data;
   * Collection of the patient's clinical history;
   * Collection of information about the history of specific pathology and comorbidities.

   Thereafter, standardized tests for psychological, neuropsychological and associated clinical conditions will be administered. In addition, there will be at least one psychoeducation meeting that can also be conducted in groups. The following tests will be administered:
   * SF 36 Questionnaire or SF 12 Questionnaire;
   * MaugerI CaRdiac preventiOn-Questionnaire (MICRO-Q);
   * Mini-mental state examnation (MMSE);
   * Beck's Depression Inventory (BDI);
   * Beck's Anxiety Inventory (BAI);
   * Zarit Burden Inventory (ZBI);
   * Eat-10 test for monitoring swallowing ability and/or Swallowing Disturbance Questionnaire (SDQ).
   * STOPBANG questionnaire and/or 2ABN3M score;
   * Voice assessment using GIRBAS Scale and VHI. Feasibility will be assessed by considering adherence to the monitoring program through testicular assessments that will be performed not only at the baseline visit (T0) but also at the six-month follow-up (T1).
2. Follow-up visit. For each patient, the assessment tests will be repeated at the same time as the periodic follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 85 years;

  * Confirmed diagnosis of cardiovascular disease;
  * Presence of chronic cardiovascular disease;
  * Absence of cognitive impairment or mild/moderate cognitive impairment (Mini Mental Score >26);
  * Patient who has given informed consent personally or through Legal Representative

Exclusion Criteria:

* - Presence of severe psychiatric and neurological disorders
* Presence of end-stage oncological disease.
* Severe visual impairment that cannot be corrected by dioptric lenses

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A minimum of 218 patients recruited from those afferent at the U.O.S.D. Cardiology with NICU P.O. "Piemonte" in Messina will participate in the survey. Statistical power analysis was performed using G*Power software for a linear regression test, assuming a slope (H1) of 0.2 with a significance level (α) of 0.05 and a power (1 - β) of 0.85. The primary outcome variable considered for the calculation was the result of the SF-12 (or SF-36) test as a summary index of the effectiveness of psychoeducation. The calculation indicated a sample of 218 subjects as adequate for the purpose of detecting the hypothesized effect
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
effectiveness of psychoeducation | 24 months
  The primary outcome variable considered for calculation is the result of the SF-12 (or SF-36) test as a summary index of the effectiveness of psychoeducation.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cappadona, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cappadona I, Ielo A, Pagano M, Anselmo A, Micali G, Giambo FM, Duca A, D'Aleo P, Costanzo D, Carcione G, Dispenzieri C, Speciale F, Bramanti P, Bramanti A, Garofano M, Corallo F. Observational protocol on neuropsychological disorders in cardiovascular disease for holistic prevention and treatment. Future Cardiol. 2025 May;21(6):349-358. doi: 10.1080/14796678.2025.2483155. Epub 2025 Mar 21. PMID 40117170